CLINICAL TRIAL: NCT03166215
Title: A Phase 1b/2a Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Escalation Study With an Open-Label Part to Examine the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TAK-935 as an Adjunctive Therapy in Subjects With Developmental and/or Epileptic Encephalopathies
Brief Title: Study of TAK-935 as an Adjunctive Therapy in Participants With Developmental and/or Epileptic Encephalopathies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Healx AI (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-935-2001; U1111-1192-7890 (Other: WHO)
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Results first posted 2020-01-10 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Developmental and/or Epileptic Encephalopathies
Keywords: Drug therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Placebo (Placebo Comparator): TAK-935 matching-placebo tablets, orally or through gastrostomy tube (G-tube)/ percutaneous endoscopic gastrostomy (PEG) tube, twice daily (BID) from Days 1 to 30 in dose titration period.
  Interventions: Drug: TAK-935
- Part 1: TAK-935 (Experimental): TAK-935 100 mg, tablet, orally or through G-tube/PEG tube, BID from Days 1 to 10 followed by TAK-935 100 mg tablets x2, orally or through G-tube/PEG tube, BID from Days 11 to 20 followed by TAK-935 100 mg tablets x3, orally or through G-tube/PEG tube, BID from Days 21 to 30 in dose titration period. The dose of TAK-935 was escalated or de-escalated during Part 1 as per investigator's discretion.
  Interventions: Drug: Placebo
- Part 2: TAK-935 (Experimental): TAK-935 100 mg tablets x2, orally or through G-tube/PEG tube, BID from Days 31 to 40 followed by TAK-935 100 mg tablets x1, x2 or x3, orally or through G-tube/PEG tube, BID from Days 31 to Day 85 as per investigator's discretion in the maintenance period. At the end of Part 2, the dose of TAK-935 was de-escalated until discontinuation.
  Interventions: Drug: TAK-935

INTERVENTIONS:
Drug: TAK-935 — TAK-935 tablets.
  Arms: Part 1: Placebo; Part 2: TAK-935
Drug: Placebo — TAK-935 placebo-matching tablets.
  Arms: Part 1: TAK-935

SUMMARY:
The purpose of this study is to characterize the multiple-dose safety and tolerability profile of TAK-935 in adult participants with developmental and/or epileptic encephalopathies.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-935. TAK-935 is being tested to treat people who have developmental and/or epileptic encephalopathies. This study will look at safety, tolerability and pharmacokinetics of people who take TAK-935. Study drug will be administered in a double-blind manner in Part 1 and in an open-label manner in Part 2.

The study will enroll approximately 20 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups in Part 1-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* TAK-935
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient

Participants will receive placebo or 100 milligram (mg) TAK-935 tablets, orally or through stable G-tube/PEG tube, BID, in Part 1 (Day 1) and dose will be increased to 200 mg (Day 11) BID and to 300 mg (Day 21) BID in dose titration period. All participants who complete the Double-Blind Treatment Period in Part 1 will have the option to continue directly into the Open-Label Treatment Period in Part 2 where they will receive TAK-935 as two 100 mg tablets (total dose is 200 mg TAK-935) orally or through G-tube/PEG tube, BID and dose will be increased to three 100 mg tablets (total dose is 300 mg TAK-935), orally, BID (Day 41). This dose level will be maintained until the final visit (Day 85) for the dose de-escalation phase.

This multi-center trial will be conducted in North America. The overall time to participate in this study is 121 days excluding screening period of 30-41 days. Participants will make multiple visits to the clinic, and a follow-up phone call will be conducted on Day 91 and at the end of the 30-day follow-up period (Day 121), participants will return to the clinic for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has a documented clinical diagnosis of developmental and/or epileptic encephalopathies with countable bilateral motor seizures, defined as an average of greater than or equal to (>=) 2 per month during the past 3 months, based on the investigator's assessment, and a monthly average of >=1 per month during the Baseline Period, based on the seizure diary record.
2. Has been taking 1 to 4 antiepileptic drug (AEDs) at a stable dose for >=4 weeks before Screening and the participant or participant's legally acceptable representative is willing to keep the regimen(s) stable throughout the study.
3. Has an average of >=1 bilateral motor seizure per month during the 4-week Baseline Period (that is., drop seizures, tonic-clonic, tonic, bilateral clonic, atonic, myoclonic-atonic, myoclonic-tonic-clonic, focal seizures with bilateral hyperkinetic motor features).
4. Must agree to not post any participant's personal medical data related to the study or information related to the study on any web site or social media site (example, Facebook, Twitter) until the study has been completed.
5. For participants with G-tube/PEG tube, G-tubes/PEG tubes should have been placed and been functioning for at least 3 months prior to screening. Naso-gastric tubes are not allowed.

Exclusion Criteria:

1. Has received TAK-935 in a previous clinical study or as a therapeutic agent.
2. Was admitted to a medical facility for treatment of status epilepticus requiring mechanical respiration within 3 months before Screening.
3. Had a vagal nerve stimulator implanted within 6 months before Screening and settings have been changed within 1 month of the Screening Visit and/or anticipated to change during the study.
4. Is on ketogenic diet that has been started within 6 months of the Screening Visit, has been changed within 1 month of the Screening Visit, or is anticipated to change during the study.
5. Has degenerative eye disease.
6. Has a history of suicidal behavior or any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening. If the participant is unable to comply with the C-SSRS due to developmental status, a parent proxy may be used for the completion of the C-SSRS. The Investigator may also use clinical judgment, which must then be documented in the source document.
7. Positive for human immunodeficiency virus, hepatitis B, or hepatitis C infections. (Note that participants who have been vaccinated against hepatitis B [hepatitis B surface antibody (Ab)-positive] who are negative for other markers of prior hepatitis B infection [example, negative for hepatitis B core Ab] are eligible. Also note that participants who are positive for hepatitis C Ab are eligible as long as they have a negative hepatitis C viral load by quantitative polymerase chain reaction [qPCR]).
8. Has an abnormal and clinically significant ECG at Screening in the opinion of the investigator, for example, second or third degree heart block or a corrected QT interval (QTc) greater than (>) 450 millisecond (msec). Entry of any participant with an abnormal but not clinically significant ECG must be approved and documented by signature by the principal investigator or appropriately qualified delegate.
9. Has abnormal clinical laboratory test results at Screening that suggest a clinically significant underlying disease. If the participant has alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2.5*the upper limit of normal (ULN), the Medical Monitor should be consulted.
10. Has received any excluded medications, procedures, or treatments during the time periods.
11. Has any a history of alcohol, opioid, or other drug use disorder, as per the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, within the previous 2 years before Screening. Medical marijuana use is allowed.
12. Has unstable, clinically significant neurologic (other than the disease being studied), psychiatric, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, hematopoietic, or endocrine disease or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor Clinical Science, Study Director — Takeda
Locations (11):
- United States (11):
  - Xenoscience, Phoenix, Arizona
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - University of South Florida, Tampa, Florida
  - Center for Integrative Rare Disease Research, Atlanta, Georgia
  - Bluegrass Epilepsy Research, Lexington, Kentucky
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - The Comprehensive Epilepsy Care Center for Children and Adults, St Louis, Missouri
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Virginia Health Sciences Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Halford JJ, Sperling MR, Arkilo D, Asgharnejad M, Zinger C, Xu R, During M, French JA. A phase 1b/2a study of soticlestat as adjunctive therapy in participants with developmental and/or epileptic encephalopathies. Epilepsy Res. 2021 Aug;174:106646. doi: 10.1016/j.eplepsyres.2021.106646. Epub 2021 Apr 22. PMID 33940389

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 investigative sites in the United States from 17 August 2017 to 19 September 2018.
Pre-assignment Details: Participants with a diagnosis of developmental and/or epileptic encephalopathies were enrolled to receive TAK-935 or placebo in Part 1 [Double Blind Treatment Period (TP)] and Part 2 (Open Label TP).
Groups:
- Part 1: Placebo: TAK-935 matching-placebo tablets, orally or through gastrostomy tube (G-tube)/percutaneous endoscopic gastrostomy (PEG) tube, twice daily (BID) from Days 1 to 30 in dose titration period.
Period: Part 1 (Double-blind TP: Days 1 - 30)
Arm/Group | Part 1: Placebo | Part 1: TAK-935 | Part 2: TAK-935
Started | 4 | 14 | 0
Completed | 4 | 12 | 0
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 0
Period: Part 2 (Open-Label TP: Days 31 - 85)
Arm/Group | Part 1: Placebo | Part 1: TAK-935 | Part 2: TAK-935
Started | 0 | 0 | 16
Completed | 0 | 0 | 14
Not Completed | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Randomized set included all participants who were randomly assigned to treatment through the interactive voice response system/ interactive web response system (IVRS/IWRS).
Groups:
- Part 1: Placebo: TAK-935 matching-placebo tablets, orally or through G-tube/PEG tube, BID from Days 1 to 30 in dose titration period.
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: TAK-935 | Total
Number analyzed (Participants) | 4 | 14 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (8.38) | 29.4 (7.83) | 29.1 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 4 | 10 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 4 | 12 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 13 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 14 | 18
Height [Mean (Standard Deviation); unit: cm] | 170.78 (14.115) | 163.80 (9.746) | 165.35 (10.802)
Weight [Mean (Standard Deviation); unit: kg] | 86.35 (26.651) | 68.57 (21.702) | 72.52 (23.310)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is participants weight in kilograms (kg) divided by his or her height in meters squared (m^2).
  kg/m^2 | 29.08 (5.688) | 24.61 (6.639) | 25.61 (6.562)
Epilepsy Diagnosis [Count of Participants; unit: Participants] — GDD is Global Developmental Delay.
  Participants
    Cerebral Dysgenesis | 0 | 1 | 1
    Complex Partial Seizure Disorder | 0 | 1 | 1
    Dravet Syndrome | 0 | 1 | 1
    Epilepsy | 1 | 2 | 3
    Epileptic Encephalopathy | 1 | 3 | 4
    Frontal Lobe Epilepsy | 0 | 1 | 1
    Hypothalamic Hamartoma | 0 | 1 | 1
    Infantile Spasms | 0 | 1 | 1
    Infantile Spasms That Went On To Lennox-Gastaut | 0 | 1 | 1
    Lennox-Gastaut Syndrome | 1 | 4 | 5
    Medically Intractable Focal Epilepsy | 0 | 1 | 1
    Mental Retardation | 0 | 2 | 2
    Partial Seizures With Secondary Generalization | 0 | 1 | 1
    Epilepsy With Significant Learning Problem and GDD | 1 | 0 | 1
    Tuberous Sclerosis | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Treatment-Emergent Adverse Event (TEAE), as Reported by the Participants or Participant's Caregivers or Observed by the Investigator, After TAK-935 Treatment
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug
Time Frame: From first dose up to 30 days post last dose (approximately up to 120 days)
Population: Safety Analysis Set for Parts 1 and 2 included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Placebo | Part 1: TAK-935 | Part 2: TAK-935
Number analyzed (Participants) | 4 | 14 | 16
percentage of participants | 100 | 71.4 | 68.8

2. Secondary Outcome: Drug Clearance (CL) and Intercompartmental Clearance (Q) for TAK-935 Calculated Using the Observed Value of the Last Quantifiable Concentration
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 5 hours) post-dose; Days 11 and 21 pre-dose and 1-hour post-dose; Days 31, 41, and 85 pre-dose
Population: Pharmacokinetic (PK) Analysis Set for Parts 1 and 2 included all participants who received at least 1 dose of study drug and have at least 1 post-dose measurable TAK-935 or metabolite of TAK-935 (M-I) plasma concentration.
Measure: Mean (Standard Deviation); unit: L/hr
Groups:
- TAK-935 100 mg BID: TAK-935 100 mg, tablet, orally or through G-tube/PEG tube, BID for 10 days in Part 1 and for 44 days in Part 2.
- TAK-935 200 mg BID: TAK-935 100 mg tablets x2, orally or through G-tube/PEG tube, BID for 10 days in Part 1 and Part 2.
- TAK-935 300 mg BID: TAK-935 100 mg tablets x3, orally or through G-tube/PEG tube, BID for 10 days in Part 1 and for 44 days in Part 2.
Arm/Group | TAK-935 100 mg BID | TAK-935 200 mg BID | TAK-935 300 mg BID
Number analyzed (Participants) | 13 | 16 | 13
L/hr
  CL | 259.4 (148.1) | 195.8 (116.3) | 190 (108.5)
  Q | 100.6 (22.24) | 70.99 (14.6) | 57.77 (11.36)

3. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Central Compartment (Vc) and Peripheral Compartment (Vp) for TAK-935 Calculated Using the Observed Value of the Last Quantifiable Concentration
Time Frame: as for outcome 2
Population: PK Analysis Set for Parts 1 and 2 included all participants who received at least 1 dose of study drug and have at least 1 post-dose measurable TAK-935 or M-I plasma concentration.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | TAK-935 100 mg BID | TAK-935 200 mg BID | TAK-935 300 mg BID
Number analyzed (Participants) | 13 | 16 | 13
L
  Vc | 56.59 (22.72) | 60.51 (23.79) | 62 (26.54)
  Vp | 677.1 (296.2) | 474.3 (201.9) | 352.9 (138.7)

4. Secondary Outcome: Absorption Rate Constant (Ka) for TAK-935
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | TAK-935 100 mg BID | TAK-935 200 mg BID | TAK-935 300 mg BID
Number analyzed (Participants) | 13 | 16 | 13
1/hr | 2.13 (0) | 2.13 (0) | 2.13 (0)

5. Secondary Outcome: Cmax,ss: Maximum Observed Plasma Concentration for TAK-935 at Steady State
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-935 100 mg BID | TAK-935 200 mg BID | TAK-935 300 mg BID
Number analyzed (Participants) | 13 | 16 | 13
ng/mL | 269.6 (159.6) | 639.8 (354.8) | 975.3 (411.5)

6. Secondary Outcome: AUC0-tau,ss: Area Under the Plasma Concentration-time Curve Over the Dosing Interval for TAK-935 at Steady State
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-935 100 mg BID | TAK-935 200 mg BID | TAK-935 300 mg BID
Number analyzed (Participants) | 13 | 16 | 13
ng*hr/mL | 562.5 (406.8) | 1437 (909) | 2188 (1357)

7. Secondary Outcome: Cav,ss: Average Plasma Concentration During a Dosing Interval at Steady State for TAK-935
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-935 100 mg BID | TAK-935 200 mg BID | TAK-935 300 mg BID
Number analyzed (Participants) | 13 | 16 | 13
ng/mL | 46.9 (33.9) | 119.8 (75.75) | 182.3 (113.1)

8. Secondary Outcome: Ctrough,ss: Plasma Concentration Immediately Prior to Dosing for TAK-935 at Steady State
Time Frame: Days 1, 11, 21; Days 31, 41 and 85 pre-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-935 100 mg BID | TAK-935 200 mg BID | TAK-935 300 mg BID
Number analyzed (Participants) | 13 | 16 | 13
ng/mL | 10.5 (13.83) | 26 (29.2) | 30.2 (29.12)

9. Secondary Outcome: Percentage of Participants With at Least 1 Markedly Abnormal Value for Clinical Laboratory Evaluations After TAK-935
Description: Clinical Laboratory parameters: hematology, serum chemistry and urinalysis. Participants with at least 1 markedly abnormal values during treatment period were reported: Erythrocytes: <0.8xLLN->1.5xULN, Hematocrit: <0.8x LLN >1.2xULN,Hemoglobin: <0.8xLLN->1.2xULN Leukocytes: <0.5xLLN, Platelets (10^9/L): <75x10^9/L->600x10^9/L, Prothrombin Ratio: >1.5xULN, Alanine Aminotransferase: >3xULN, Albumin:<25 g/L, Alkaline Phosphatase: >3xULN,Alpha-1 Acid Glycoprotein: <47 mg/DL->125 mg/DL, Aspartate Aminotransferase:>3xULN, Bicarbonate:<8.0 mmol/L, Calcium:<1.75 mmol/L->2.88 mmol/L, Chloride:<75 mmol/L->126 mmol/L, Cholesterol: >7.72,Creatine Kinase:>5xULN, Creatinine:>177 umol/L, Gamma Glutamyl Transferase: >3xULN, Glucose:<2.8 mmol/L- >19.4 mmol/L,HDL Cholesterol: <1.04 mmol/L->1.55 mmol/L, LDL Cholesterol: <1.30 mmol/L->4.14 mmol/L, Potassium:<3.0 mmol/L->6.0 mEq/L, Protein:<0.8xLLN->1.2 x ULN, Sodium: <130 mmol/L->150 mmol/L, Triglycerides: >2.5xULN, Urea Nitrogen: >10.7 mmol/L.
Time Frame: From first dose up to last dose (up to Day 85)
Population: Safety Analysis Set for Parts 1 and 2 included all participants who received at least 1 dose of study drug. Data reported is the data available for the specific parameter.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Placebo | Part 1: TAK-935 | Part 2: TAK-935
Number analyzed (Participants) | 4 | 14 | 16
percentage of participants
  Alpha-1 Acid Glycoprotein (>125 mg/DL): number analyzed (Participants) | 4 | 9 | 14
  Alpha-1 Acid Glycoprotein (>125 mg/DL) | 0 | 11.1 | 14.3
  Gamma Glutamyl Transferase ( >3 x ULN): number analyzed (Participants) | 4 | 11 | 15
  Gamma Glutamyl Transferase ( >3 x ULN) | 0 | 9.1 | 6.7
  HDL Cholesterol (<1.04 mmol/L): number analyzed (Participants) | 4 | 11 | 16
  HDL Cholesterol (<1.04 mmol/L) | 75.0 | 18.2 | 40.0
  HDL Cholesterol (>1.55 mmol/L): number analyzed (Participants) | 4 | 11 | 15
  HDL Cholesterol (>1.55 mmol/L) | 0 | 27.3 | 13.3
  LDL Cholesterol (>4.14 mmol/L): number analyzed (Participants) | 4 | 11 | 16
  LDL Cholesterol (>4.14 mmol/L) | 0 | 9.1 | 0
  Potassium (>6.0 mmol/L): number analyzed (Participants) | 4 | 11 | 16
  Potassium (>6.0 mmol/L) | 0 | 9.1 | 0

10. Secondary Outcome: Percentage of Participants With at Least 1 Markedly Abnormal Value for Vital Signs After TAK-935
Description: Vital signs included heart rate, blood pressure and body temperature. markedly abnormal values during treatment period were categorized as: heart rate 1,3 and 5 min standing (beats/min) <50->120, systolic blood pressure 1,3 and 5 min standing (mmHg) <85->180, diastolic blood pressure 1,3 and 5 min standing (mmHg) <50->110 and body temperature (degree centigrade) <35.6- >37.7. Only categories with values have been reported.
Time Frame: From first dose up to 30 days post last dose (approximately up 120 days)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Placebo | Part 1: TAK-935 | Part 2: TAK-935
Number analyzed (Participants) | 4 | 14 | 16
percentage of participants
  Diastolic Blood Pressure 3 min Standing (<50 mmHg): number analyzed (Participants) | 3 | 7 | 8
  Diastolic Blood Pressure 3 min Standing (<50 mmHg) | 33.3 | 0 | 0
  Diastolic Blood Pressure 5 min Sitting (<50 mmHg) | 0 | 7.1 | 0
  Diastolic Blood Pressure 5 min Supine (<50 mmHg): number analyzed (Participants) | 4 | 9 | 16
  Diastolic Blood Pressure 5 min Supine (<50 mmHg) | 25.0 | 0 | 0
  Heart Rate 1 min Standing (>120 beats/min): number analyzed (Participants) | 3 | 6 | 8
  Heart Rate 1 min Standing (>120 beats/min) | 0 | 16.7 | 0
  Heart Rate 5 min Sitting (<50 beats/min) | 50.0 | 0 | 6.3
  Heart Rate 5 min Supine (<50 beats/min): number analyzed (Participants) | 4 | 9 | 16
  Heart Rate 5 min Supine (<50 beats/min) | 25.0 | 0 | 0
  Systolic Blood Pressure 5 min Sitting (<85 mmHg) | 0 | 7.1 | 0
  Temperature (<35.6 C): number analyzed (Participants) | 4 | 13 | 16
  Temperature (<35.6 C) | 25.0 | 7.7 | 18.8

11. Secondary Outcome: Percentage of Participants With at Least 1 Markedly Abnormal Value for Electrocardiogram (ECG) Parameters After TAK-935
Description: A 12-lead ECG was performed. Markedly abnormal values during treatment period were categorized as: ECG ventricular rate <50->120, PR Interval, (msec) <=80->=200, QRS Duration, (msec) <=80->=180, QT Interval, (msec) <=50->=460, QTcF Interval, (msec) <=50->=500 OR >=30 change from baseline and >=450 milliseconds, RR interval <600->=1440.
Time Frame: From first dose up to last dose (up to Day 85)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Placebo | Part 1: TAK-935 | Part 2: TAK-935
Number analyzed (Participants) | 4 | 14 | 16
percentage of participants
  ECG Ventricular Rate (<50 beats/min): number analyzed (Participants) | 3 | 8 | 16
  ECG Ventricular Rate (<50 beats/min) | 33.3 | 0 | 0
  QRS Duration (<=80 msec): number analyzed (Participants) | 3 | 8 | 15
  QRS Duration (<=80 msec) | 0 | 12.5 | 6.7
  RR Interval (<=600 msec): number analyzed (Participants) | 3 | 8 | 15
  RR Interval (<=600 msec) | 0 | 0 | 13.3

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days post last dose (approximately up to 120 days)
Arm/Group | Part 1: Placebo | Part 1: TAK-935 | Part 2: TAK-935
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/14 | 3/16
Other Adverse Events (participants affected / at risk) | 4/4 | 10/14 | 11/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=4) | Part 1: TAK-935 (N=14) | Part 2: TAK-935 (N=16)
Seizure Cluster (Nervous system disorders) | 0 | 1 | 2
Seizure (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=4) | Part 1: TAK-935 (N=14) | Part 2: TAK-935 (N=16)
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 3
Agitation (Psychiatric disorders) | 0 | 1 | 1
Communication disorder (Psychiatric disorders) | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1 | 0
Listless (Psychiatric disorders) | 0 | 0 | 1
Sleep talking (Psychiatric disorders) | 1 | 0 | 0
Tic (Psychiatric disorders) | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 3 | 0
Headache (Nervous system disorders) | 1 | 2 | 0
Lethargy (Nervous system disorders) | 0 | 2 | 2
Seizure (Nervous system disorders) | 0 | 0 | 3
Balance disorder (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 0
Repetitive speech (Nervous system disorders) | 0 | 1 | 0
Sedation (Nervous system disorders) | 1 | 0 | 0
Tonic convulsion (Nervous system disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 0
Pyrexia (General disorders) | 0 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Human bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT03166215/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT03166215/SAP_001.pdf